CLINICAL TRIAL: NCT04321460
Title: Multicentre, Double-blind, Randomized, Placebo-controlled, Parallel-group Efficacy and Safety Study of LRG-002 Hard Capsules (Lek d.d., Slovenia) Used in the Prophylaxis of Antibiotic-associated Diarrhea in Adults.
Brief Title: Study of LRG-002 Hard Capsules (Lek d.d., Slovenia) Used in the Prophylaxis of Antibiotic-associated Diarrhea in Adults.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT_002_LRG_CAP
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-12

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRG-002 (Experimental): LRG-002 once daily for 14 days
  Interventions: Drug: LRG-002
- Placebo (Placebo Comparator): Placebo once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LRG-002 — Capsules containing live lyophilized probiotic bacteria of Lactobacillus genus
  Arms: LRG-002
Drug: Placebo — Capsules containing placebo
  Arms: Placebo

SUMMARY:
The goal of this study was to investigate the efficacy and safety of LRG-002 investigational medicinal product, capsules (Lek d.d., Slovenia) in comparison with placebo, as an adjunct treatment for prophylaxis of antibiotic-associated diarrhea (AAD) in patients with acute respiratory diseases (ARDs) receiving a standard antimicrobial therapy.

DETAILED DESCRIPTION:
This study was the prospective, multi-centered, double-blinded, randomized, parallel-group clinical study. The study investigated the efficacy and safety of LRG-002 investigational medicinal product, capsules (Lek d.d., Slovenia) in comparison with placebo, as an adjunct treatment for prophylaxis of antibiotic-associated diarrhea (AAD) in patients with acute respiratory diseases (ARDs) receiving a standard antimicrobial therapy.

The study comprised the following periods:

Study Periods Visit 1 (Day 1): Screening + randomization + initiation of treatment

Patients started participating in the study after signing the Informed Consent Form. Having completed screening tests, eligible patients were randomized on the same day to receive either LRG-002 or matching placebo capsules, each as an adjunct to the prescribed antibiotic. The treatment group was determined by randomization at a center ratio. Study subjects were supplied with the patient diary and blinded investigational product (investigational medicinal product or placebo) depending on the assigned treatment group. Patients could start study treatment only after receiving appropriate training. On Day 1, the study started in both groups from randomization and administration of the first dose of the investigational product depending on the assigned group after randomization:

Group T, treated with LRG-002: a single dose of 1 oral hard capsule taken during meals with some water; the product was to be taken orally 2 times per day for 14 days.

Group R, provided with placebo:a single dose of 1 oral hard capsule taken during meals with some water; the product is to be taken orally 2 times per day for 14 days.

Visit 2 (Day 7): Intermediate Follow-up Visit

Visit 3 (Day 15) : Visit 3 was scheduled at Day 15 when a patient was to come to the study site bringing along the completed diary, unused laboratory kit, unused product and empty packages.

ELIGIBILITY:
Patients will be considered eligible for study participation if they meet the following inclusion criteria:

1. An Informed Consent Form for study participation voluntarily signed by a patient;
2. Male and female subjects, 18 to 65 years of age inclusive;
3. Antibacterial treatment for active ARDs started/to be started on the first day of the study (7-day course of oral beta-lactam antibiotic). Only one AB should be used per subject, in an outpatient setting. Diagnostic procedures of ARD and the prescription of antibiotic therapy should be completed before signing of the Informed Consent Form.
4. Female patients will be considered as eligible for study participation if they are: Unable to become pregnant or Capable of childbirth, but with negative pregnancy test at the screening visit, and the patient agrees to continuously and properly use one a following suitable methods of contraception Male participants,. together with their partner, are to use appropriate contraception during the entire study period starting from signing of the Informed Consent Form and until the study end, and for 30 days after study completion;

6. The ability to understand the information about the clinical study, readiness to comply with the study protocol requirements, ability to take the investigational products and evaluate symptoms on his (or her) own using diary/questionnaires as per protocol; 7. Ability to maintain the habitual lifestyle throughout the study, including diet. 8. Willing not to consume any products containing probiotics during participation in the clinical trial. 9. Willing not to take part in any other study during the present trial.

Patients will not be eligible for study enrollment if they have one or more of the following criteria:

1. Any therapy (including medications, medical devices and dietary supplements) that can influence the stool consistency, according to the Investigator's opinion, should not be used within 14 days prior to Visit 1;
2. Use of immunosuppressive, immunostimulating and immunomodulating agents including drugs of herbal origin and dietary supplements within 30 days prior to the study start;
3. Use of anti-rejection medication after stem cell or solid organ transplant;
4. Use of systemic glucocorticosteroids within 8 weeks prior to the study start;
5. Use of proton pump inhibitors within 3 months prior to Visit 1;
6. Chemotherapy or radiation;
7. History of recurrent diarrhea;
8. Patient has diarrhea or loose stool within 2 days prior to the study start;
9. Patient has severe ARD expected to require an administration of antibiotics therapy for more than 7 days or prescription of additional antibiotics;
10. Use of antimicrobials within 3 months prior to the study start;
11. Use of yeast/probiotic/fermented products within 2 weeks prior to the first visit;
12. Known allergy/hypersensitivity to the investigational medicinal product in the medical history;
13. Immunocompromised patients;
14. Known digestion/absorption disorders of the gastrointestinal tract (e.g. inflammatory bowel disease, celiacia, pancreatitis, motility disorders etc.) and/or gastrointestinal surgery;
15. Known irritable bowel syndrome;
16. Known small intestinal bacterial overgrowth;
17. Patient has pyrexia of more than 38°C;
18. Pregnant and/or breastfeeding women;
19. Participation in other clinical trials of medicinal products or medical devices at the screening Visit or within 30 days before the screening Visit;
20. Surgical intervention within 30 days before the screening visit or planned surgical treatment during the trial (before a follow-up visit is completed), including diagnostic procedures or inpatient stay;
21. Known or suspected alcohol and/or drug addiction;
22. A suspected low compliance or incapability of the patient to perform the procedures and comply with restrictions according to the trial protocol (e.g., due to mental disorders);
23. Potential for translocation of probiotic across bowel wall (Presence of an active bowel leak, acute abdomen, active intestinal disease including colitis, or significant bowel dysfunction; presence of neutropenia or anticipation of neutropenia after chemotherapy; radiation therapy);
24. Any disorders of cardiovascular, renal, hepatic, gastrointestinal, endocrine and nervous systems, or other conditions/diseases which, in the Investigator's opinion, may render study participation unsafe for a patient or may affect a test result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Sandoz Investigative Site, Moscow
  - Sandoz Investigative Site, Nizhny Novgorod
  - Sandoz Investigative Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 15 sites in the Russian Federation.
Pre-assignment Details: Participants were randomized in 1:1 ratio to two arms (Treatment and Placebo).
Period: Overall Study
Arm/Group | LRG-002 | Placebo
Started | 260 | 260
Intention to Treat (ITT) Population | 260 | 260
Per-protocol (PP) Population | 252 | 248
Completed | 259 | 259
Not Completed | 1 | 1
Not completed — Participants who had no defecation or no data about it | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LRG-002 | Placebo | Total
Number analyzed (Participants) | 260 | 260 | 520
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.62 (12.93) | 41.65 (12.74) | 41.13 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 167 | 309
  Male | 118 | 93 | 211
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 259 | 259 | 518
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Occurrence of Antibiotic-associated Diarrhea (AAD) - Per Protocol (PP) Population
Description: Diarrhea is defined as loose or watery stool (Type 5-7 according to Bristol Stool Form Scale (BSFS)), three times a day (frequent bowel movements with formed stool is not considered as diarrhea) in accordance with WHO criteria; based on the diary data (BSFS) and confirmation of AAD by the investigator. BSFS scale includes Types 1 to 7 where Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicate lack of dietary fiber, and 6 and 7 indicate diarrhea. AAD (antibiotic-associated diarrhea) is defined as diarrhea associated with the antibiotic use caused by C. difficile or of otherwise not identified etiology, upon analysis of stool samples and differential diagnostics according to investigator's judgment. Diarrhea was assessed in a diary.
Time Frame: 14 days
Population: The per protocol (PP) population included all randomized participants who completed participation in the study in accordance with the protocol (have completed the prescribed period of treatment and follow-up without significant deviations from the protocol)
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 252 | 248
Participants | 4 | 17
Statistical Analysis 1: Comparison: LRG-002 vs Placebo; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 4.564, 95% CI 2-sided [1.66 to 16.039]

2. Primary Outcome: Number of Participants With the Occurrence of Antibiotic-associated Diarrhea (AAD) - Intention to Treat (ITT) Population
Description: as for outcome 1
Time Frame: 14 days
Population: The intention-to-treat (ITT) population included all randomized participants who received at least one dose of the investigational medicinal product/placebo and have completed at least one visit aimed at the evaluation of efficacy parameters (i.e., at least all the procedures of Visit 1)
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 260 | 260
Participants | 5 | 22
Statistical Analysis 1: Comparison: LRG-002 vs Placebo; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 4.716, 95% CI 2-sided [1.898 to 14.268]

3. Secondary Outcome: Mean Number of Bowel Movements Per Day
Description: Bowel movements were assessed based on the data of patient's diary
Time Frame: 14 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of bowel movements per day
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 259 | 259
Number of bowel movements per day | 1.54 (0.64) | 1.76 (0.72)

4. Secondary Outcome: Number of Participants With the Occurrence of Any Diarrhea
Description: as for outcome 1
Time Frame: 14 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 260 | 260
Participants | 6 | 23

5. Secondary Outcome: Number of Participants With the Occurrence of C. Difficile-associated Antibiotic-associated Diarrhea (AAD)
Description: as for outcome 1
Time Frame: 14 Days
Population: The intention-to-treat (ITT) population included all participants with available data, who received any study drug and had Antibiotic-associated diarrhea (AAD)
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 5 | 22
Participants | 0 | 1

6. Secondary Outcome: Number of Participants With the Occurrence of Non-C. Difficile-associated AAD
Description: Incidence of non-C. difficile-associated AAD assessed based on the data of stool analysis
Time Frame: 14 Days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 5 | 22
Participants | 5 | 21

7. Secondary Outcome: Mean Duration of Antibiotic-associated Diarrhea (AAD)
Description: AAD is defined as diarrhea associated with the antibiotic use caused by C. difficile or of otherwise not identified etiology, upon analysis of stool samples and differential diagnostics according to investigator's judgment.The duration of AAD was the time from the onset of AAD to the normalization of stool form according to Bristol Stool Scale (types 1, 2, 3 and 4 where Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid) and the presence of normal stool within 48 hours was assessed based on the data of patient's diary.
Time Frame: 14 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 5 | 22
Days | 5.4 (2.3) | 6.23 (3.72)

8. Secondary Outcome: Mean Duration of Any Diarrhea
Description: Duration of any diarrhea is defined as the time from the onset of diarrhea to the normalization of stool shape according to the Bristol Stool Form Scale (BSFS) (Types 1, 2, 3, and 4) and the presence of normal stool for 48 hours). BSFS scale includes Types 1 to 7 where Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicate lack of dietary fiber, and 6 and 7 indicate diarrhea.
Time Frame: 14 days
Population: The intention-to-treat (ITT) population included all participants with available data, who received any study drug and had incidence of any diarrhea
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 6 | 23
Days | 5 (2.28) | 6.13 (3.66)

9. Secondary Outcome: Change in Stool Consistency
Description: Individual changes in the stool consistency were classified as improved / unchanged / worsened. The calculations were conducted as follows:
  1. if more than 1 observation was available for a specific day, the maximum score was taken;
  2. each subsequent day was compared to Day 1 according to the following rules:
     * variations within 3-4 points, 1-2 points, or 5-7 points were qualified as "unchanged";
     * transfer from 1-2 points or 5-7 points to 3-4 points, as well as transfer from 5-7 points to 1-2 points were qualified as "improved";
     * transfer from 3-4 points to 1-2 points or 5-7 points, as well as transfer from 1-2 points to 5-7 points were qualified as "worsened".
     Score interpretation:
  3. 1, 2 - hard stool (constipation)
  4. 3, 4 - normal value
  5. 5, 6, 7 - loose stool
Time Frame: Baseline, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14
Population: The intention-to-treat (ITT) population included participants with available Day 1 assessment data
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 206 | 214
Participants
  Day 2 Change in the stool consistency as compared to Day 1: improved | 78 | 56
  Day 2 Change in the stool consistency as compared to Day 1: unchanged | 94 | 124
  Day 2 Change in the stool consistency as compared to Day 1: worsened | 27 | 27
  Day 2 Change in the stool consistency as compared to Day 1: no data available | 7 | 7
  Day 3 Change in the stool consistency as compared to Day 1: improved | 79 | 60
  Day 3 Change in the stool consistency as compared to Day 1: unchanged | 96 | 118
  Day 3 Change in the stool consistency as compared to Day 1: worsened | 26 | 33
  Day 3 Change in the stool consistency as compared to Day 1: no data available | 5 | 3
  Day 4 Change in the stool consistency as compared to Day 1: improved | 83 | 62
  Day 4 Change in the stool consistency as compared to Day 1: unchanged | 95 | 122
  Day 4 Change in the stool consistency as compared to Day 1: worsened | 25 | 26
  Day 4 Change in the stool consistency as compared to Day 1: no data available | 3 | 4
  Day 5 Change in the stool consistency as compared to Day 1: improved | 78 | 59
  Day 5 Change in the stool consistency as compared to Day 1: unchanged | 93 | 119
  Day 5 Change in the stool consistency as compared to Day 1: worsened | 30 | 27
  Day 5 Change in the stool consistency as compared to Day 1: no data available | 5 | 9
  Day 6 Change in the stool consistency as compared to Day 1: improved | 78 | 59
  Day 6 Change in the stool consistency as compared to Day 1: unchanged | 100 | 120
  Day 6 Change in the stool consistency as compared to Day 1: worsened | 18 | 28
  Day 6 Change in the stool consistency as compared to Day 1: no data available | 10 | 7
  Day 7 Change in the stool consistency as compared to Day 1: improved | 83 | 60
  Day 7 Change in the stool consistency as compared to Day 1: unchanged | 94 | 119
  Day 7 Change in the stool consistency as compared to Day 1: worsened | 23 | 26
  Day 7 Change in the stool consistency as compared to Day 1: no data available | 6 | 9
  Day 8 Change in the stool consistency as compared to Day 1: improved | 78 | 61
  Day 8 Change in the stool consistency as compared to Day 1: unchanged | 99 | 123
  Day 8 Change in the stool consistency as compared to Day 1: worsened | 21 | 17
  Day 8 Change in the stool consistency as compared to Day 1: no data available | 8 | 13
  Day 9 Change in the stool consistency as compared to Day 1: improved | 75 | 61
  Day 9 Change in the stool consistency as compared to Day 1: unchanged | 100 | 124
  Day 9 Change in the stool consistency as compared to Day 1: worsened | 20 | 20
  Day 9 Change in the stool consistency as compared to Day 1: no data available | 11 | 9
  Day 10 Change in the stool consistency as compared to Day 1: improved | 74 | 61
  Day 10 Change in the stool consistency as compared to Day 1: unchanged | 96 | 119
  Day 10 Change in the stool consistency as compared to Day 1: worsened | 23 | 23
  Day 10 Change in the stool consistency as compared to Day 1: no data available | 13 | 11
  Day 11 Change in the stool consistency as compared to Day 1: improved | 83 | 65
  Day 11 Change in the stool consistency as compared to Day 1: unchanged | 95 | 119
  Day 11 Change in the stool consistency as compared to Day 1: worsened | 22 | 24
  Day 11 Change in the stool consistency as compared to Day 1: no data available | 6 | 6
  Day 12 Change in the stool consistency as compared to Day 1: improved | 80 | 66
  Day 12 Change in the stool consistency as compared to Day 1: unchanged | 96 | 124
  Day 12 Change in the stool consistency as compared to Day 1: worsened | 20 | 19
  Day 12 Change in the stool consistency as compared to Day 1: no data available | 10 | 5
  Day 13 Change in the stool consistency as compared to Day 1: improved | 76 | 61
  Day 13 Change in the stool consistency as compared to Day 1: unchanged | 99 | 118
  Day 13 Change in the stool consistency as compared to Day 1: worsened | 19 | 22
  Day 13 Change in the stool consistency as compared to Day 1: no data available | 12 | 13
  Day 14 Change in the stool consistency as compared to Day 1: improved | 81 | 63
  Day 14 Change in the stool consistency as compared to Day 1: unchanged | 91 | 122
  Day 14 Change in the stool consistency as compared to Day 1: worsened | 22 | 20
  Day 14 Change in the stool consistency as compared to Day 1: no data available | 12 | 9

10. Secondary Outcome: Number of Gastrointestinal Symptoms by Severity
Description: The severity of gastrointestinal symptoms, including nausea, vomiting, flatulence, abdominal pain and decreased appetite was assessed based on the data of patient's diary. Severity of symptoms was assessed based on the 5-point verbal scale [0 to 4] where 0- symptoms were absent, 4- symptoms were very severe
Time Frame: 14 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 259 | 259
Participants
  Abdominal pain, severity: 0. No manifestations | 18 | 19
  Abdominal pain, severity: 1. Mild manifestations | 29 | 36
  Abdominal pain, severity: 2. Moderate manifestations | 7 | 4
  Abdominal pain, severity: 3. Severe manifestations | 0 | 3
  Abdominal pain, severity: No data available | 205 | 197
  Flatulence, severity: 0. No manifestations | 13 | 13
  Flatulence, severity: 1. Mild manifestations | 34 | 50
  Flatulence, severity: 2. Moderate manifestations | 30 | 40
  Flatulence, severity: 3. Severe manifestations | 5 | 6
  Flatulence, severity: No data available | 177 | 150
  Vomiting, severity: 0. No manifestations | 20 | 21
  Vomiting, severity: 1. Mild manifestations | 0 | 2
  Vomiting, severity: 2. Moderate manifestations | 0 | 0
  Vomiting, severity: 3. Severe manifestations | 0 | 0
  Vomiting, severity: No data available | 239 | 236
  Decreased appetite, severity: 0. No manifestations | 11 | 5
  Decreased appetite, severity: 1. Mild manifestations | 43 | 51
  Decreased appetite, severity: 2. Moderate manifestations | 43 | 42
  Decreased appetite, severity: 3. Severe manifestations | 8 | 10
  Decreased appetite, severity: No data available | 154 | 151
  Nausea, severity: 0. No manifestations | 21 | 20
  Nausea, severity: 1. Mild manifestations | 30 | 21
  Nausea, severity: 2. Moderate manifestations | 1 | 2
  Nausea, severity: 3. Severe manifestations | 0 | 0
  Nausea, severity: No data available | 207 | 216

11. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight assessed based on the clinical data
Time Frame: Baseline, Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 259 | 257
Kg | 0.11 (1.13) | -0.17 (0.92)

12. Secondary Outcome: Number of Participants Hospitalized
Description: Hospitalization rate was assessed based on the clinical data
Time Frame: 14 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 260 | 260
Participants | 0 | 1

13. Secondary Outcome: Number of Participants Using Standard Symptomatic Therapy
Description: The number of participants using standard symptomatic therapy (as "rescue medication") to relieve symptoms of acute diarrhea were assessed based on the clinical data
Time Frame: 14 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 260 | 260
Participants | 0 | 1

14. Secondary Outcome: Number of Days of Using Standard Symptomatic Therapy
Description: The number of days of using standard symptomatic therapy (as "rescue medication") to relieve symptoms of acute diarrhea were assessed based on the clinical data
Time Frame: 14 days
Population: Included only 1 participants who was prescribed symptomatic therapy for C. difficile-associated diarrhea
Measure: Number; unit: Days
Arm/Group | LRG-002 | Placebo
Number analyzed (Participants) | 0 | 1
Days |  | NA — Participant prematurely withdrawn from the trial therefore no analysis performed due to missing data

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study i.e until visit 3 (Day 15 ± 2) which was the treatment completion / study termination visit
Description: Any signs or symptoms were collected throughout the study i.e until visit 3 (Day 15 ± 2) which was the treatment completion / study termination visit
Arm/Group | LRG-002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/260 | 0/260
Serious Adverse Events (participants affected / at risk) | 0/260 | 1/260
Other Adverse Events (participants affected / at risk) | 116/260 | 138/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LRG-002 (N=260) | Placebo (N=260)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LRG-002 (N=260) | Placebo (N=260)
Flatulence (Gastrointestinal disorders) | 65 | 90
Nausea (Gastrointestinal disorders) | 28 | 20
Abdominal pain (Gastrointestinal disorders) | 36 | 40
Diarrhea (Gastrointestinal disorders) | 6 | 24
Decreased appetite (Metabolism and nutrition disorders) | 92 | 93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT04321460/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04321460/SAP_001.pdf